CLINICAL TRIAL: NCT02138058
Title: Double Blind Controlled Trial of Topiramate for Compulsive Buying
Brief Title: Topiramate Trial for Compulsive Buying
Acronym: TFO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Hermano Tavares, Associate professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Topiramate for oniomania
Record Dates: First submitted 2014-05-12; First posted 2014-05-14 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2015-12

CONDITIONS: Compulsive Shopping
Keywords: compulsive buying, compulsive shopping, topiramate
MeSH Terms: interventions — Topiramate

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): a 12 week placebo matching tablets plus 4 sessions of a manualized cognitive restructuring intervention
  Interventions: Behavioral: Cognitive restructuring intervention
- topiramate (Experimental): a 12 week topiramate flexible dose administration plus 4 sessions of a manualized cognitive restructuring intervention
  Interventions: Drug: Topiramate; Behavioral: Cognitive restructuring intervention

INTERVENTIONS:
Drug: Topiramate
  Arms: topiramate
Behavioral: Cognitive restructuring intervention — 4 sessions of a manualized cognitive restructuring intervention for compulsive buying
  Other Names: behavioral

SUMMARY:
It is a double blind controlled study to test the hypothesis that Topiramate is more effective than placebo in the treatment of compulsive buying, during a period of 12 weeks

DETAILED DESCRIPTION:
Compulsive buying is a prevalent disorder with no approved pharmacological treatment. Previous reports suggest that topiramate could be useful in reducing impulsivity in pathological gambling and other impulse control disorders, as well as craving in substance addictions. The goal of this study was to investigate the effectiveness of topiramate combined with brief cognitive restructuring in treating compulsive buying, compared with just cognitive restructuring treatment+placebo.

ELIGIBILITY:
Inclusion Criteria:

* Match criteria for compulsive buying, according to McElroy et al. (1994), confirmed by semi-structured interview modeled after the Schedules for clinical assessment in neuropsychiatry (SCID)
* woman within fertility age have to be already practicing an acceptable contraception method and to be negative at a pregnancy test

Exclusion Criteria:

* illiteracy
* pregnancy and breastfeeding for woman
* previous history of alcohol abuse/dependence with current elevation of liver enzymes, or a present diagnosis of alcohol abuse/dependence
* past or current drug abuse/dependence, except for nicotine
* history of current or past Fifth Edition of the Diagnostic and Statistical Manual of Mental Disorders diagnosis of bipolar disorder, schizophrenia, psychosis or any neuropsychiatric condition causing cognitive impairment
* a history of suicide attempt or acute suicide risk
* severe depression indicated by a score higher than 30 at the beck depression inventory
* current participation on psychotherapy or use of pharmacological agent or experimental dispositive for compulsive buying in the past 3 months
* current use of psychotropic drugs, except benzodiazepines
* cardiovascular disease including a history of heart attack, stroke, arrhythmia, cardiac failure in the past 5 years. Uncontrolled high blood pressure.
* chronic or acute renal or liver failure, as well as Retinopathy and thyroidopathy
* a personal or family history of nephrolithiasis
* immunodeficiency
* any blood dyscrasia
* contraindication or allergy to topiramate
* history of seizures
* dont't have a phone number for contact
* live alone and don't have a person that can inform about the shopping behavior

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2015-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Yale-Brown Compulsive-Obsessive Scale Shopping Version | 12 weeks
  It is a revised version of the Yale-Brown Obsessive-Compulsive Scale (YBOCS), created to assess both the cognitive and behaviour of compulsive buying as well as to rate the severity of the problem

SECONDARY OUTCOMES:
Clinical Global Impression scale (CGI) | 12 weeks
  The CGI scale quantifies the severity of disease and the effects of treatment, as well as overall clinical improvement.
Udvalg for KliniskeUndersøgelser Side Effect Rating Scale (UKU) | 12 weeks
  It was developed to provide a comprehensive side effect rating scale with well-defined and operationalized items to assess the side effects of psychopharmacological medications.

OTHER OUTCOMES:
Social adjustment | 12 weeks
  The social Adjustment scale (SAS) is a self-report scale that assesses seven specific areas: work, social, life and leisure, extended family relationship, marital relationship, relationship with offsprings, domestic life and financial situation

CONTACTS AND LOCATIONS:
Overall Officials: Hermano Tavares, Professor, Principal Investigator — associate
Locations (1):
- Associação Viver Bem, São Paulo, São Paulo, Brazil

REFERENCES:
- See also: Non for profit organization that supports Impulse Control patients and their relatives — http://www.associacaoviverbem.org.br